CLINICAL TRIAL: NCT05688917
Title: Effect of Green Coffee Supplementation on Inflammatory Biomarkers in Obese Patients With Metabolic Syndrome
Brief Title: Green Coffee Effect on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Damanhour University (Other)
Responsible Party: Principal Investigator, Naglaa Khedr, Professor of Biochemistry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FPTU-11-2020
Record Dates: First submitted 2021-01-24; First posted 2023-01-18 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Supportive Care; Metabolic Syndrome; Obesity; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hypertension

STUDY DESIGN:
Intervention Model Description: 160 obese patients supplemented with GCBE capsules (800 mg) daily for six months
Who Masked: Participant, Investigator
Masking Description: double-blind randomised controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- green been extract treated group (Experimental): Participants included in the study were maintained on a balanced diet and supplemented with Green Coffee Bean (Coffea Arabica) extract capsules (800 mg/capsule
  Interventions: Dietary Supplement: Green coffee been extract
- Placebo group (Placebo Comparator): Participants included in the study were maintained on a balanced diet and supplemented with placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Green coffee been extract — supportive treatment
  Arms: green been extract treated group
Other: Placebo — Placebo capsule
  Arms: Placebo group

SUMMARY:
The present study aimed to investigate the effect of green coffee bean extract (GCBE) on the inflammatory biomarkers in obese patients with a metabolic syndrome via analyzing some inflammatory biomarkers as resistin, TNF-α, total sialic acid, homocysteine, high sensitivity C-reactive protein (hs-CRP) and anti-inflammatory cytokine, adiponectin

DETAILED DESCRIPTION:
160 obese patients supplemented with either GCBE capsules (800 mg) daily or placebo for 6 months and advised to take a balanced diet. Blood samples were collected at baseline and after three months of supplementation

ELIGIBILITY:
Inclusion Criteria:

Participants were enrolled if they were

* aged 20-60y
* waist circumference >102 cm in male; 88 cm in female
* triglycerides ≥150 mg/dL (1.7 mmol/L)
* HDL-C<40 mg/dL (1.03 mmol/L) in males & <50 mg/dL (1.29 mmol/L) in females
* systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg.

Exclusion Criteria:

* liver, kidney, coronary artery disease, type I diabetes, autoimmune diseases, cancer, infection, smoking, recent major surgery, routine coffee consumption, pregnancy or breast-feeding, use of anti-inflammatory drugs, corticosteroids, hormone replacement therapy, weight-loss and anti-hypercholesterolemic medications three months or less prior to enrolment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Adiponectin (µg/mL) | six months
  Serum Level
TNF-α (pg/mL) | six months
  Serum Level
Resistin (ng/mL) | six months
  Serum Level
Homocysteine (µmol/L) | six months
  Serum Level
Hs-CRP (mg/L) | Six months
  Serum Level

SECONDARY OUTCOMES:
BMI (kg/m2) | six months
  Weight / hight squared.
LDL-C (mg/dL) | six Months
  calculated according to Friedewald formula.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass. Prof., Study Chair — Damanhour University
Locations (1):
- Naglaa Khedr, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Not applicable. the data will published in specialized journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: data after analysis

REFERENCES:
- [Background] Lange E, Keszycka PK, Palkowska-Gozdzik E, Billing-Marczak K. Comparison of Glycemic Response to Carbohydrate Meals without or with a Plant-Based Formula of Kidney Bean Extract, White Mulberry Leaf Extract, and Green Coffee Extract in Individuals with Abdominal Obesity. Int J Environ Res Public Health. 2022 Sep 25;19(19):12117. doi: 10.3390/ijerph191912117. PMID 36231426
- [Result] Roshan H, Nikpayam O, Sedaghat M, Sohrab G. Effects of green coffee extract supplementation on anthropometric indices, glycaemic control, blood pressure, lipid profile, insulin resistance and appetite in patients with the metabolic syndrome: a randomised clinical trial. Br J Nutr. 2018 Feb;119(3):250-258. doi: 10.1017/S0007114517003439. Epub 2018 Jan 8. PMID 29307310
- [Result] Meshkani M, Saedisomeolia A, Yekaninejad M, Mousavi SA, Ildarabadi A, Vahid-Dastjerdi M. The Effect of Green Coffee Supplementation on Lipid Profile, Glycemic Indices, Inflammatory Biomarkers and Anthropometric Indices in Iranian Women With Polycystic Ovary Syndrome: A Randomized Clinical Trial. Clin Nutr Res. 2022 Oct 28;11(4):241-254. doi: 10.7762/cnr.2022.11.4.241. eCollection 2022 Oct. PMID 36381474
- [Derived] Khedr NF, Zahran ES, Ebeid AM, Melek ST, Werida RH. Effect of green coffee on miR-133a, miR-155 and inflammatory biomarkers in obese individuals. Diabetol Metab Syndr. 2024 Oct 28;16(1):256. doi: 10.1186/s13098-024-01478-7. PMID 39468643